CLINICAL TRIAL: NCT02771106
Title: Neuroimaging and Neurovision Rehabilitation of Oculomotor Dysfunction in Mild Traumatic Brain Injury
Status: Completed | Type: Observational
Sponsor: Hennepin Healthcare Research Institute (Other)
Collaborators: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: HSR #13-3702
Record Dates: First submitted 2016-05-02; First posted 2016-05-12 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Traumatic Brain Injury; Vision Difficulty
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- vision dysfunction: This group are subjects with mild TBI who have been diagnosed with profound oculomotor (vision) dysfunction per objective measurements taken by the HCMC developmental optometrist. These subjects will undergo neuro vision rehabilitation.
  Interventions: Other: neuro vision rehabilitation
- control: This group are subjects with mild TBI who have no oculomotor (vision) dysfunction per objective measurements taken by the HCMC developmental optometrist

INTERVENTIONS:
Other: neuro vision rehabilitation — Neuro vision rehabilitation used to treat vision dysfunction following TBI
  Groups: vision dysfunction

SUMMARY:
Mild TBI subjects will initially be identified by providers in the Hennepin County Medical Center (HCMC) TBI Clinic. The subjects will then undergo objective testing by the developmental optometrist to confirm if they do or do not have vision dysfunction related to the mTBI. At the Center of Magnetic Resonance Research (CMRR) located at the University of Minnesota (U of M), the whole brain will be imaged using resting state and task functional MRI and diffuse tensor imaging (DTI) using a high field 3 Tesla (T) MRI. The subjects will then receive neurovision rehabilitation if they are in the vision dysfunction group. This treatment is standard care. Both groups will then undergo repeat objective vision testing by the developmental optometrist at 3 and 6 months to confirm that vision dysfunction has resolved. Resting state and task fMRI and DTI will be done at the same time to compare functional and structural connectivity changes between the 2 groups.

DETAILED DESCRIPTION:
The primary objectives are: 1) To localize changes following mild traumatic brain injury (mTBI) in subjects with vision dysfunction using functional magnetic resonance imaging (fMRI) and diffusion tensor imaging (DTI). 2) To demonstrate the effectiveness of neuro vision rehabilitation (NVR) on vision dysfunction initiated within nine months following mTBI by normalizing objective visual measurements as well as changes on fMRI and DTI.

Mild (TBI) comprises 80% of the 3.65 million brain injuries in the United States and costs an estimated 17 billion dollars annually. Mild TBI is a challenging diagnosis and can be as disabling as a severe TBI when chronic symptoms develop. In the past several years, researchers have found that a somewhat silent majority of mTBI patients who develop lasting symptoms have concurrent vision dysfunction. This cohort of patients with post-traumatic visual difficulty, regardless of mechanism of injury, seem to demonstrate more significant and lasting disability and poorer overall outcome than other TBI cohorts, yet these correlations have not been adequately studied. The studies that have been performed have found that visual dysfunctions may not spontaneously improve and become chronic in absence of direct diagnosis and treatment. Time after injury has been shown in studies to have no influence on incidence or frequency of visual difficulties but once identified, these pervasive visual dysfunctions significantly improve in response to interventions such as prescription glasses and NVR.

For the past 16 months, the Center for Magnetic Resonance Research (CMRR) at the University of Minnesota (U of M) and the TBI Center at the Hennepin County Medical Center (HCMC) have closely collaborated in a pilot study. The goal of this study was to identify the location in the brain of post traumatic visual changes in acute mTBI subjects (< 9 months from injury date, ages 18-55) using resting state and task fMRI and DTI. Mild TBI subjects who had vision dysfunction (vision group) were compared to mTBI subjects who did not have any vision difficulties (controls). Task fMRI imaging demonstrated significant decreased brain activity in the vision dysfunction subjects as compared to the controls in certain key vision areas. Diffusion tensor imaging showed significant changes in certain areas of the corpus callosum.

This trial is designed as a longitudinal clinical study. Fifteen mTBI patients with vision dysfunction (vision group) fitting the inclusion/exclusion criteria and 15 patients with mTBI but with no findings on the visual screen (control group) within 9 months of their injury will be included in the study. No subject will be excluded on the basis of sex/gender, race or ethnicity. These mTBI subjects will initially be identified by physicians in the HCMC TBI Clinic. If agreeable, consent will be obtained at both HCMC as well as prior to their baseline MRI scans at CMRR. The subjects will then undergo objective testing by a specialized eye doctor at HCMC to confirm if they do or do not have vision dysfunction related to the mTBI. At CMRR, within 2 weeks of the visual testing, the whole brain will be imaged using resting state and task fMRI and DTI using a 3T MRI machine. The subjects will then receive neurovision rehabilitation for approximately 3 months at HCMC if they are in the vision group. This treatment is standard care for this population. Both groups will then undergo repeat objective vision testing by the specialized eye doctor at 3 and 6 months to confirm that vision dysfunction has resolved. Resting state and task fMRI and DTI will be done at the same time to compare functional and structural connectivity changes between the 2 groups.

Mild TBI is a significant cause of disability especially when symptoms become chronic. In HCMC's clinical experience, this chronicity is often linked to vision difficulties. Vision dysfunction will continue until properly identified and treated, especially with neuro vision rehabilitation. The goals of this research study are to better understand cerebral structural and metabolic changes associated with as well as the effectiveness of neuro vision rehabilitation on post traumatic vision dysfunction by utilizing resting state and task fMRI and DTI. A positive outcome will have a significant impact on the diagnosis and care of the considerable numbers of mTBI patients suffering from vision dysfunction, especially because neurovision rehabilitation will be more utilized by the medical community. In turn, the overall functional outcomes after mTBI will improve, greatly relieving the suffering and disability for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Mild TBI (GCS score > 13), Post Traumatic Amnesia < 24 hours, no brain CT findings
* Diagnosed with vision dysfunction by developmental optometrist
* Age equal to or > 16 years- 55 years.
* Injury between 1 - 9 months
* Informed consent obtained

Exclusion Criteria:

* Any type of bio-implant activated by mechanical, electronic, or magnetic means
* Any type of ferromagnetic bio-implant that could potentially be displaced
* Pregnant females
* Significant anxiety and/or claustrophobia
* Subjects who cannot adhere to the experimental protocol
* Brain tumor or stroke or severe traumatic brain injury or history of severe mental retardation
* Any chemotherapy, immunomodulatory agents, or radiation treatment affecting the brain
* Two or more seizures, or been given a diagnosis of epilepsy
* Known ocular problems including orbital fractures, monocular vision, strabismus, - Lasik surgery for monofixation, cataracts with visual acuity > 20/40
* History of intractable migraines
* History of major psychiatric disorder
* Taking medications which interfere with visual process
* Taking illicit drugs such as marijuana, cocaine, heroin, etc
* Age < 16 and > 55 years
* GCS score < 13
* Current TBI or still symptomatic from prior mTBI > 9 months
* Any vision rehabilitation
* Near point convergence > 70 cm or sustained diplopia
* Cranial nerve II, III, IV, or VI palsy
* Any findings on clinical brain CT or MRI
* Any subject with a professional or academic link to the PI

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects who have suffered a mild traumatic brain injury who fit the below inclusion/exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2020-08-21 (Actual); Study Completion 2020-08-21 (Actual)

PRIMARY OUTCOMES:
To localize changes following mild traumatic brain injury in subjects with vision dysfunction using magnetic resonance imaging (MRI). | 18 months
2) The effectiveness of neuro vision rehabilitation on vision dysfunction initiated within nine months following mTBI will be shown using magnetic resonance imaging by comparing aggregate data of 15 vision dysfunction subjects to 15 control subjects. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Sarah B Rockswold, MD, Principal Investigator — Minneapols Medical Research Foundation
Locations (1):
- Hennepin County Medical Cetner, Minneapolis, Minnesota, United States